CLINICAL TRIAL: NCT03868592
Title: Long-term, Substantial Weight Loss and Insulin Regulation of Lipolysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael D. Jensen, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-005349
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Study insulin action and adipose function before and after weight loss from gastric sleeve surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastric sleeve surgery (Experimental): before and after weight loss from bariatric surgery
  Interventions: Procedure: Gastric sleeve/bariatric surgery

INTERVENTIONS:
Procedure: Gastric sleeve/bariatric surgery — weight loss

SUMMARY:
It is not known how much improvement in insulin regulated lipolysis (the breakdown of triglycerides) occurs following substantial, sustained weight loss. Researchers will test the effects of inflammation and lipolysis regulation in people before and after bariatric surgery (sleeve gastrectomy) to answer these questions.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the adipose inflammatory cell and cytokine content in Class III obesity is related to lipolysis insulin resistance and, if so, whether sustained, substantial weight loss one year following bariatric surgery reduces inflammation in parallel with improved insulin regulation of lipolysis

ELIGIBILITY:
Inclusion Criteria:

* BMI 40 - 50 kg/m2.
* Mo active physical illness that would interfere with mobility or weight loss after bariatric surgery

Exclusion Criteria:

* Type 1 or Type 2 Diabetes diagnosis or fasting plasma glucose ≥126 mg/dL
* Active coronary artery disease
* Participation in structured exercise (>2 times per week for 30 minutes or longer)
* Smoking
* Medications known to affect adipose tissue metabolism (e.g., beta blockers, corticosteroids)
* Renal insufficiency (serum creatinine > 1.5mg/dl)
* Chronic active liver disease (Bilirubin > 17mmol/L, AST > 144 IU/L, or ALT>165IU/L)
* Pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
adipose macrophage content, adipose IL-6 and TNF gene expression | Before bariatric surgery and approximately 1 year after surgery
  Adipose tissue macrophage content as assessed by immunohistochemistry using stains for CD36, CD14 and CD206 will be done. mRNA expression for IL-6 and TNF will be measured
insulin regulation of lipolysis (IC50) | Before bariatric surgery and approximately 1 year after surgery
  The ability of insulin to suppress FFA palmitate release will be assessed using a 2-step insulin clamp and isotope dilution techniques for palmitate kinetics

SECONDARY OUTCOMES:
adipocyte perilipin 1 and HSL and ATGL | Before bariatric surgery and approximately 1 year after surgery
  These proteins will be measured using capillary Western methods.

OTHER OUTCOMES:
Long-term, substantial weight loss and insulin regulation of lipolysis | 1 year
  Patients will undergo studies of insulin regulation of FFA release combined with adipose biopsies before and one year after bariatric surgery (gastric sleeve). We will relate the improvement in insulin-regulation of lipolysis to changes in adipose tissue lipolysis proteins as measured by changes in adipocyte perilipin 1 dephosphorylation in response to insulin.
Long-term, substantial weight loss and insulin regulation of lipolysis | 1 year
  Patients will undergo studies of insulin regulation of FFA release combined with adipose biopsies before and one year after bariatric surgery (gastric sleeve). We will relate the improvement in insulin-regulation of lipolysis to changes in adipose tissue lipolysis proteins as measured by changes in adipocyte HSL dephosphorylation in response to insulin.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Jensen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No